CLINICAL TRIAL: NCT07366294
Title: Effects of Lemongrass (Cymbopogon Citratus) on Nicotine Dependence, Cotinine Levels, and Related Biomarkers in Adult Smokers
Brief Title: Lemongrass (Cymbopogon Citratus) on Nicotine Dependence, Cotinine Levels, and Related Biomarkers in Adult Smokers
Acronym: CCIVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Titin Andri Wihastuti (Other)
Collaborators: University of Brawijaya (Other)
Responsible Party: Sponsor-Investigator, Titin Andri Wihastuti, Principal Investigator (Professor), University of Brawijaya
Organization: University of Brawijaya (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00147.3/UN10.A0501/B/2024; 00147.3/UN10.A0501/B/PT01.03.2 (Other: Universitas Brawijaya)
Record Dates: First submitted 2026-01-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Nicotine Dependence; Cigarette Smoking; Tobacco Use Disorder; Psychological Stress; Sleep Disturbance
Keywords: Cymbopogon citratus; Nicotine Dependence; Smoking Biomarkers; Oxidative Stress; Adult Smokers
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Stress, Psychological; Parasomnias

STUDY DESIGN:
Intervention Model Description: Participants are allocated in parallel to receive either a lemongrass (Cymbopogon citratus) inhaler and vapor intervention or a control condition, with outcomes assessed concurrently across study arms.
Masking Description: This study is conducted as an open-label trial. Participants, care providers, investigators, and outcome assessors, including laboratory analysts, are aware of the assigned intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants in this arm do not receive lemongrass inhaler or liquid vapor. They continue their usual smoking behavior and daily activities without any additional intervention for the duration of the study.
- Lemongrass Inhaler (Experimental): Participants receive a lemongrass (Cymbopogon citratus) inhaler administered by inhalation according to the study protocol.
  Interventions: Other: Lemongrass Inhaler
- Lemongrass Liquid Vapor (Experimental): Participants receive lemongrass (Cymbopogon citratus) liquid vapor administered via vaporization according to the study protocol.
  Interventions: Other: Lemongrass Liquid Vapor
- Lemongrass Inhaler and Liquid Vapor (Experimental): Participants receive a combination of lemongrass (Cymbopogon citratus) inhaler and liquid vapor administered concurrently according to the study protocol.
  Interventions: Other: Lemongrass Inhaler and Liquid Vapor

INTERVENTIONS:
Other: Lemongrass Inhaler — Participants receive a lemongrass (Cymbopogon citratus) inhaler administered by inhalation according to the study protocol.
  Arms: Lemongrass Inhaler
Other: Lemongrass Liquid Vapor — Participants receive lemongrass (Cymbopogon citratus) liquid vapor administered via vaporization according to the study protocol.
  Arms: Lemongrass Liquid Vapor
Other: Lemongrass Inhaler and Liquid Vapor — Participants receive a combination of lemongrass (Cymbopogon citratus) inhaler and liquid vapor administered concurrently according to the study protocol.
  Arms: Lemongrass Inhaler and Liquid Vapor

SUMMARY:
The goal of this clinical trial is to learn whether lemongrass (Cymbopogon citratus) inhaler and liquid vapor interventions affect nicotine dependence and related biological and behavioral outcomes in adult smokers. The study will also evaluate changes in blood biomarkers, psychological well-being, and lifestyle-related measures. The main questions it aims to answer are:

* Do lemongrass inhalers and/or liquid vapor reduce nicotine dependence and cotinine levels in adult smokers?
* How do these interventions affect blood lipid profile and biomarkers of inflammation, oxidative stress, endothelial function, and stress response, including interleukin-6 (IL-6), malondialdehyde (MDA), superoxide dismutase (SOD), nitric oxide (NO), cortisol, and nicotinic acetylcholine receptors (nAChRs)?
* Do lemongrass inhaler and liquid vapor influence appetite, physical fitness, sleep quality, and psychological status measured using the Depression, Anxiety, and Stress Scale (DASS)?

Researchers will compare participants receiving lemongrass inhaler, lemongrass liquid vapor, or a combination of both to a control group receiving no intervention to evaluate the effects of the interventions.

Participants will:

* Receive a lemongrass inhaler, lemongrass liquid vapor, a combination of both, or no intervention according to group assignment
* Continue their usual daily activities during the study period
* Provide blood samples and complete questionnaires to assess biochemical markers, nicotine dependence, appetite, fitness level, sleep quality, and psychological status

DETAILED DESCRIPTION:
Cigarette smoking is associated with nicotine dependence and a wide range of biological, psychological, and lifestyle-related alterations, including oxidative stress, inflammation, neuroendocrine dysregulation, and impaired functional well-being. Complementary inhalation-based approaches using plant-derived aromatic compounds may offer supportive benefits by modulating smoking-related biological and behavioral responses.

This open-label, parallel-group interventional study is conducted to evaluate the effects of lemongrass (Cymbopogon citratus)-based inhaler and liquid vapor formulations in adult smokers. Participants are assigned to receive a lemongrass inhaler, lemongrass liquid vapor, a combination of both interventions, or no intervention. The study is designed to compare intervention groups with a non-intervention control group under real-world conditions.

The lemongrass inhaler and vapor products are formulated to provide consistent aromatic exposure and have undergone standardized physical, organoleptic, and stability evaluations prior to use. Interventions are administered according to predefined study procedures.

The study assesses biological, behavioral, and functional responses related to smoking exposure and dependence, including biochemical, neuroendocrine, and psychosocial domains. Data are collected using standardized laboratory methods and validated assessment tools.

By integrating objective biomarkers with behavioral and functional measures, this study aims to provide insight into the potential role of lemongrass-based inhalation interventions as supportive strategies for addressing smoking-related health effects in adult smokers.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 30 years
* Current cigarette smokers reporting consumption of ≥5 cigarettes per day
* Moderate to high nicotine dependence, defined as a Fagerström Test for Nicotine Dependence (FTND) score≥5
* Members of the academic community of the Faculty of Health Sciences, Universitas Brawijaya, Malang, East Java, Indonesia
* Willing and able to provide informed consent and comply with study procedures

Exclusion Criteria:

* Current use of smoking cessation medications
* History of lemongrass allergy
* Presence of chronic respiratory conditions
* History of severe cardiovascular disease
* History of severe psychiatric disorders
* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Change in Nicotine Dependence (FTND Score) | Baseline up to 4 weeks
  Change in nicotine dependence measured using the Fagerström Test for Nicotine Dependence (FTND), a validated 6-item questionnaire with total scores ranging from 0 to 10, where higher scores indicate greater nicotine dependence.

SECONDARY OUTCOMES:
Change in Cotinine Levels | Baseline up to 4 weeks
  Change in blood cotinine concentration measured using enzyme-linked immunosorbent assay (ELISA), reported in nanograms per milliliter (ng/mL).
Change in Lipid Profile | Baseline up to 4 weeks
  Change in blood lipid profile parameters, including total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, and triglycerides, measured using standard enzymatic laboratory methods and reported in milligrams per deciliter (mg/dL).
Change in Inflammatory and Oxidative Stress Biomarkers | Baseline up to 4 weeks
  Change in interleukin-6 concentration measured using ELISA and reported in picograms per milliliter (pg/mL), malondialdehyde concentration reported in nanomoles per milliliter (nmol/mL), superoxide dismutase activity reported in units per milliliter (U/mL), and nitric oxide concentration reported in micromoles per liter (µmol/L).
Change in Neuroendocrine and Receptor-Related Biomarkers | Baseline up to 4 weeks
  Change in cortisol concentration measured using ELISA and reported in micrograms per deciliter (µg/dL), and nicotinic acetylcholine receptor-related measures assessed using laboratory-based immunoassays and reported in relative expression units.
Change in Appetite | Baseline up to 4 weeks
  Change in appetite assessed using a standardized appetite questionnaire, reported as a total score ranging from 0 to 10, where higher scores indicate greater appetite.
Change in Sleep Quality | Baseline up to 4 weeks
  Change in sleep quality assessed using a validated sleep questionnaire, reported as a total score ranging from 0 to 10, where higher scores indicate poorer sleep quality.
Change in Psychological Status | Baseline up to 4 weeks
  The Depression, Anxiety, and Stress Scale (DASS) consists of three subscales with score ranges of 0-42 for each subscale, where higher scores indicate greater severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Titin A Wihastuti, Professor, Principal Investigator — Brawijaya University
Locations (1):
- University of Brawijaya, Malang, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to confidentiality concerns, small sample size, and the absence of participant consent and infrastructure for secure data sharing. Study findings will be reported in aggregate form.

REFERENCES:
- [Background] Moreira da Silva TL, Beltrame FL, Ferrari PC. Lemongrass essential oil micro- and nanoencapsulation for industrial application: Production techniques and potential applications. Arch Pharm (Weinheim). 2024 Jun;357(6):e2300726. doi: 10.1002/ardp.202300726. Epub 2024 Mar 28. PMID 38548681
- [Background] Adhikary K, Banerjee P, Barman S, Bandyopadhyay B, Bagchi D. Nutritional Aspects, Chemistry Profile, Extraction Techniques of Lemongrass Essential Oil and It's Physiological Benefits. J Am Nutr Assoc. 2024 Feb;43(2):183-200. doi: 10.1080/27697061.2023.2245435. Epub 2023 Aug 14. PMID 37579058
- [Background] Rabbani A, Khaliq A, Mudgil P, Maqsood S, Nazir A. Recent Advances in Lemongrass Essential Oil: Food Safety, Preservation, and Bioactivity in Food Systems. Compr Rev Food Sci Food Saf. 2026 Jan;25(1):e70350. doi: 10.1111/1541-4337.70350. PMID 41347276